CLINICAL TRIAL: NCT05025085
Title: A Phase 1 Study Investigating AGEN1777 as a Single-Agent and in Combination With a PD-1 Inhibitor in Patients With Advanced Solid Tumors
Brief Title: A Study Investigating AGEN1777 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA115-P01; C-1400-01 (Other: Agenus Inc.)
Record Dates: First submitted 2021-08-10; First posted 2021-08-27 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer
Keywords: Solid Tumors; Dose Escalation; Monotherapy; Combination Therapy; Anti-PD-1; Undisclosed Target

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy with AGEN1777 (Experimental): 3+3 Dose escalation of AGEN1777 will be administered by Intravenous (IV) infusion every 3 weeks (each cycle is 21 days [3 weeks]).
  Interventions: Drug: AGEN1777
- AGEN1777 in combination with a PD-1 inhibitor (Experimental): 3+3 Dose escalation of AGEN1777 in combination with a PD-1 inhibitor will be administered by IV infusion with specified dose on specified days.
  Interventions: Drug: AGEN1777; Drug: a PD-1 inhibitor

INTERVENTIONS:
Drug: AGEN1777 — An immunoglobulin gamma (IgG1) antibody
Drug: a PD-1 inhibitor — Anti-programmed cell death protein 1 (Anti-PD-1) antibody monoclonal antibody
  Arms: AGEN1777 in combination with a PD-1 inhibitor

SUMMARY:
This study is a multicenter, Phase 1 study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of AGEN1777 as a single agent and when used in combination with a PD-1 inhibitor in participants with advanced, metastatic solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced solid tumor for which no acceptable standard therapy available or progressed on or after standard therapies.
2. Measurable disease on baseline imaging based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
3. Life expectancy of at least 3 months and an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

1. Active infection requiring treatment.
2. Lack of recovery for participants who had major surgical procedure within 4 weeks prior to first dose of protocol therapy.
3. Clinically significant cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
4. Corrected QT interval (QTc) (corrected for heart rate using Fridericia's formula prolongation) >480 msec at screening except for right bundle branch block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLT) of AGEN1777 as a Single-Agent and in Combination with a PD-1 inhibitor | Day 1 through Day 21
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to 2 years and 90 days

SECONDARY OUTCOMES:
Maximum Observed Concentration at Steady State (Cmax-ss) of Serum AGEN1777 and a PD-1 inhibitor | Day 1 Up to End of Treatment (up to 2 years)
Serum AGEN1777 Anti-Drug Antibody (ADA) Determination | Day 1 of Cycle 1 (Cycle = 21 days) through Day 1 of Cycle 5. Incidence of ADA
Serum a PD-1 inhibitor Anti-Drug Antibody (ADA) Determination | Day 1 Up to End of Treatment (up to 2 years)
Complete Response (CR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) Based on Investigator's assessment | From Day 1 of Cycle 1 (each cycle is 21 days [3 weeks]) until every 9 weeks (±7 days) for 12 months, and every 12 weeks (±7 days) thereafter up to 2 years or until progressive disease or unacceptable toxicity
Partial Response (PR) per RECIST v1.1 Based on Investigator's Assessment | From Day 1 of Cycle 1 (each cycle is 21 days [3 weeks]) until every 9 weeks (±7 days) for 12 months, and every 12 weeks (±7 days) thereafter up to 2 years or until progressive disease or unacceptable toxicity
Duration of Response (DOR) per RECIST v1.1 Based on Investigator's Assessment | From Day 1 of Cycle 1 (each cycle is 21 days [3 weeks]) until every 9 weeks (±7 days) for 12 months, and every 12 weeks (±7 days) thereafter up to 2 years or until progressive disease or unacceptable toxicity.
Stable Disease (SD) per RECIST v1.1 Based on Investigator's Assessment | From Day 1 of Cycle 1 (each cycle is 21 days [3 weeks]) until every 9 weeks (±7 days) for 12 months, and every 12 weeks (±7 days) thereafter up to 2 years or until progressive disease or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - Local Institution - 165, Grand Rapids, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Local Institution - 024, Southfield, Michigan
  - Local Institution - 072, Cincinnati, Ohio
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Local Institution - 0001, Providence, Rhode Island
  - Local Institution - 164, Dallas, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center Thoracic-Head & Neck Med Onc, Houston, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html